CLINICAL TRIAL: NCT02574234
Title: Influence of Apelin Levels on Postoperative Cognitive Disorders After Orthopedic Surgery in Elderlies
Brief Title: Influence of Apelin Levels on Postoperative Cognitive Disorders After Orthopedic Surgery in Elderlies (APOCOGNIT)
Acronym: APOCOGNIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/14/7313
Record Dates: First submitted 2015-08-26; First posted 2015-10-12 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Delirium
Keywords: Postoperative cognitive disorders POCD; inflammation; Surgery
MeSH Terms: conditions — Delirium; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with orthopedic surgery (Experimental): Patients will be included in the consultation of anesthesia. The usual laboratory tests will be carried out and a determination of apelin and inflammatory cytokines. Assessment of cognitive functions using the Informant Questionnaire on Cognitive Decline in the Elderly (ICQODE), Mini Mental State examination (MMS) and the scale of Instrumental activities of daily living (IADL).
  Day of surgery: liquid sampling cerebrospinal. Day 1 to day 7 postoperatively: determination of inflammatory cytokines and apelin, postoperative delirium research (Confusion Assessment Method (CAM)), residual cognitive dysfunction research (MMS, IADL, IQCODE).
  3 months after operation: evaluation of cognitive performance (IQCODE, IADL)
  Interventions: Other: Determination of apelin and inflammatory cytokines; Other: Assessment of cognitive functions; Other: Liquid sampling cerebrospinal; Other: Postoperative delirium research; Other: Residual cognitive dysfunction research

INTERVENTIONS:
Other: Determination of apelin and inflammatory cytokines — A blood sample will be conducted at baseline, on day 1 and day 7 post operative to meter inflammatory cytokines (IL1B, IL1-ra, IL6) and apelin.
Other: Assessment of cognitive functions — Evaluation of preoperative cognitive performance by achieving a IQCODE, an MMS and an IADL scale.
Other: Liquid sampling cerebrospinal — Determination of the concentrations of inflammatory cytokines and apelin in cerebrospinal fluid perioperatively.
Other: Postoperative delirium research — Using the scale Confusion Assessment Method (CAM) for screening and delirium diagnosis. This research will be daily lasted, during the first 7 days postoperative.
Other: Residual cognitive dysfunction research — Evaluation of postoperative cognitive performance by achieving a IQCODE, an MMS and an IADL scale realised on day 1 and day 7 postoperative. Realization of the IQCODE and IADL three months after the operation in a telephone interview.

SUMMARY:
No successful strategy is proposed to patients submitted to important surgery to reduce the incidence of postoperative cognitive disorders (POCD) onset. This project propose to measure plasma levels of apelin in wide population submitted to orthopedic surgery. Apelin could be involved in anti-inflammatory processes. Apelin levels before and after surgery correlated to postoperative cognitive disorders symptom measured by PET-Scan could be an important predictive or diagnostic marker to adapt therapeutic strategy to fight against postoperative cognitive disorders.

DETAILED DESCRIPTION:
It has been now clearly shown that important surgery with general anesthesia could be strongly associated to postoperative cognitive disorders few months after the intervention especially in elderlies. No strategy is really efficient to fight against this phenomenon that could lead to Alzheimer disease development. In order to prognosticate and characterize the potential risk to develop cognitive troubles after a surgery, this study propose to evaluate the potential predictive capacity of apelin in a cohort of young and old adult undergoing an orthopedic surgery. Apelin is a peptide involved in different physiological as well physiopathological pathways. This peptide, involved in osteogenesis and inflammatory processes, has also been described to be neuroprotective. Yet, hippocampic neuroinflammation has been related in case of postoperative cognitive disorders in human as well as in mice model of surgery. Taken together, these results seem to indicate that apelin could be a therapeutic target and be predictive of the postoperative cognitive disorders onset.

This study will measure plasma apelin levels in young and old adult one day before and after a programed orthopedic surgery. Moreover, to correlate apelin amounts with inflammation processes, protocol will quantify inflammatory cytokines in plasma (IL6, IL1, TNFα). These results will be compared to measures of brain b-amyloid deposit assessed by PET-Scan technology.

The follow-up of the patients will be done during 3 months in order to evaluate the postoperative cognitive disorders or the cognitive troubles associated to surgery (memory fail, decrease of cognitive reserve…).

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to a programed orthopedic surgery
* Patients with pre- and post-surgery check-up.

Exclusion Criteria:

* Non programed orthopedic surgery (emergency)
* Patients with sepsis
* Patients submitted to orthopedic surgery but with ambulatory management.
* Existence of justice backup, curators or supervision.
* Absence of indication for a pre- or post-surgery check-up.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium occurrence. | day1 to day 7 post-operation
  Evaluation of the occurrence of postoperative delirium evaluated by the Confusion Assessment Method (CAM)

SECONDARY OUTCOMES:
Evaluation of postoperative cognitive functions. | day 1 to day 7 and 3 month after post-operation
  Evaluation with IQCODE questionary (Informant Questionary on Cognitive Decline in the Elderly)
Assessment of the autonomy. | day 1 to day 7 and 3 month after post-operation
  Evaluation with IADL scale (Instrumental Activities Scale of Everyday Life)
Plasma concentration of apelin. | day 1 to day 7 post operation
Plasma concentration of inflammatory cytokines. | 24 hours before operation, day 1 to day 7 post operation
Concentration of inflammatory cytokines and apelin in the cerebrospinal fluid. | day 0 (operation day)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent MINVILLE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, service d'orthopédie et traumatologie, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverstein JH, Timberger M, Reich DL, Uysal S. Central nervous system dysfunction after noncardiac surgery and anesthesia in the elderly. Anesthesiology. 2007 Mar;106(3):622-8. doi: 10.1097/00000542-200703000-00026. No abstract available. PMID 17325520
- [Background] Deiner S, Silverstein JH. Postoperative delirium and cognitive dysfunction. Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i41-46. doi: 10.1093/bja/aep291. PMID 20007989
- [Background] Price CC, Garvan CW, Monk TG. Type and severity of cognitive decline in older adults after noncardiac surgery. Anesthesiology. 2008 Jan;108(1):8-17. doi: 10.1097/01.anes.0000296072.02527.18. PMID 18156877
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Cibelli M, Fidalgo AR, Terrando N, Ma D, Monaco C, Feldmann M, Takata M, Lever IJ, Nanchahal J, Fanselow MS, Maze M. Role of interleukin-1beta in postoperative cognitive dysfunction. Ann Neurol. 2010 Sep;68(3):360-8. doi: 10.1002/ana.22082. PMID 20818791
- [Result] Labaste F, Delort F, Ferre F, Bounes F, Reina N, Valet P, Dray C, Minville V. Postoperative delirium is a risk factor of institutionalization after hip fracture: an observational cohort study. Front Med (Lausanne). 2023 Aug 15;10:1165734. doi: 10.3389/fmed.2023.1165734. eCollection 2023. PMID 37649978